CLINICAL TRIAL: NCT00593294
Title: Comparison of Oral Contraceptive Versus Physical Exercise Effects on Cardiovascular and Metabolic Risk Factors in PCOS Women
Brief Title: Oral Contraceptive and Cardiovascular Risk in PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Francesco Orio, Dpt of Mol and Clin Endocrinology and Oncology Federico II University of Naples
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-12-2871; CE209/07
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2007-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; oral contraceptives; physical exercise; CVR
MeSH Terms: conditions — Polycystic Ovary Syndrome; Motor Activity | interventions — Exercise; Ethinyl Estradiol; Vitamins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A,1,I (Experimental)
  Interventions: Behavioral: Physical exercise
- B, 2, II (Active Comparator)
  Interventions: Drug: OC - Drospirenone plus Ethynylestradiol
- C,3,III (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin, polyvitamins tablets

INTERVENTIONS:
Behavioral: Physical exercise — 45 minutes each day for three times/week for 6 months
  Arms: A,1,I
Drug: OC - Drospirenone plus Ethynylestradiol — 1 cp for 21 days each month for 6 months of OC (Drospirenone 3 mg plus Ethynylestradiol 30 microgram = Yasmin, Schering, Milan, Italy)
  Arms: B, 2, II
Dietary Supplement: Vitamin, polyvitamins tablets — Tablet of vitamin 1cp for 21 days each month for 6 months
  Arms: C,3,III

SUMMARY:
Oral contraceptive therapy is routinely used for the treatment of menstrual disturbances of patients with polycystic ovary syndrome (PCOS).

To date, the cardiovascular risk (CVR) of the oral contraceptives (OC) are known but no data are available on the CVR in PCOS patients treated with OC or physical exercise.

The purpose of this study is to compare the effects of OC to physical exercise on the CVR of PCOS women and show the hormonal and metabolic effects of these two different treatment.

We hypothesize that physical exercise has the same beneficial effects of OC therapy on hormonal and metabolic features of PCOS women with less cardiovascular consequences.

DETAILED DESCRIPTION:
One hundred and fifty PCOS women will be enrolled. The diagnosis of PCOS was made based according to the Rotterdam criteria (1). Specifically, patients with anovulation and clinical and/or biochemical hyperandrogenism were enrolled.

Patients will be randomly allocated in three groups (OC, physical exercise and placebo group) using a computer-software. Fifty PCOS patients will be treated with OC (Drospirenone 3 mg, Ethynylestradiol 30 microgram = Yasmin, Schering, Milan,Italy) other fifty PCOS will be undergone physical exercise, whereas other fifty will be treated with placebo tablets (one tablet once daily; placebo group). The duration of the treatment will be 6 months.

Patients treated with OC will be instructed to follow their usual diet and physical activity, whereas patients undergone to physical exercise will be instructed to follow a detailed regular physical training program and for the diet they will be advised for the quality of food to eat. All subjects will be nonsmokers and none will drink alcoholic beverages.

Each subject will undergo follow-up visits under (at three and 6 months from treatment starting) and after treatment (at three and 6 months from treatment withdrawal). At each follow-up visit, in all subjects the same operator will perform clinical, hormonal, metabolic and cardiovascular assessments by carotid and brachial artery US

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome

Exclusion Criteria:

* Age <18 or >40 years
* BMI higher than 30 and lower than 18
* Pregnancy
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, nonclassical congenital adrenal hyperplasia, use of OC, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic or antiobesity drugs or other hormonal drugs within the previous 6 months
* Subjects with neoplastic, metabolic (including glucose intolerance), hepatic, and cardiovascular disorder or other concurrent medical illness (i.e. diabetes, renal disease, or malabsorptive disorders, cephalea)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes: Intima media thickness by carotid ultrasonography (US) and Flow Mediated Dilation by brachial artery US | Basal and after 3 and 6 months

SECONDARY OUTCOMES:
Secondary Outcomes: Clinical, hormonal, and metabolic assessments | Basal and after 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Orio, MD,PhD, Principal Investigator — Department of Molecular and Clinical Endocrinology and Oncology University Federico II Naples Italy; Gaetano Lombardi, MD, Study Director — Department of Molecular and Clinical Endocrinology and Oncology University Federico II Naples Italy; Stefano Palomba, MD, Study Chair — Chair of Obstetrics and Gynecology, University "Magna Graecia" Catanzaro, Italy
Locations (1):
- Department of Molecular and Clinical Endocrinology and Oncology, University "Federico II", Naples, Naples, Italy

REFERENCES:
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538